CLINICAL TRIAL: NCT05270694
Title: Understanding Factors Influencing COVID-19 Testing and Vaccination in Immigrant, Low-income and Unhoused Populations, and Testing Targeted Interventions [3U54GM115516=04S2 RADx-UP]
Brief Title: Evaluating Public Health Interventions to Improve COVID-19 Testing Among Underserved Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathleen Fairfield (Other)
Collaborators: MaineHealth (Other)
Responsible Party: Sponsor-Investigator, Kathleen Fairfield, Physician Scientist, and Associate Professor of Medicine, Public Health & Community Medicine at Tufts University School of Medicine, MaineHealth
Organization: MaineHealth (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1795294
Record Dates: First submitted 2022-02-09; First posted 2022-03-08 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: COVID-19 testing; Low-income populations; Immigrant populations; Unhoused populations; Uninsured populations
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: 150 participants will be enrolled into the cohort, with 15 participants from each of the 10 specific populations of interest (3 groups that access different health services for low-income/uninsured, unhoused individuals, and 6 different immigrant groups)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 Testing (Experimental): The cohort participants will attend an in-person training on how to take an at-home COVID-19 test and also be provided with five at-home test kits at the training and every other month for a total of 35 kits over the course of a year.
  Interventions: Behavioral: Public Health Intervention Package

INTERVENTIONS:
Behavioral: Public Health Intervention Package — The intervention package consists of two components:
  1. At the time of study enrollment, participants will attend an in-person training on how to properly take an at-home COVID-19 test. Study staff will verbally walk through the steps of the test with the participant while the participant administers the test on themselves, with the opportunity to ask questions and receive corrective feedback, as needed.
  2. To make COVID-19 testing more accessible, participants will be provided five at-home COVID-19 testing kits at the training and then every other month throughout the course of the year-long study for a total of 35 kits.

SUMMARY:
The COVID-19 pandemic has disproportionately affected people from underserved and vulnerable populations such as low-income/uninsured, unhoused, and immigrant communities. These populations in the US are at a higher risk of acquiring COVID-19 because of poverty, type of occupation, greater use of public transit, living in multigenerational housing, lack of access to quality healthcare, and more. Despite greater risk of being infected and dying of COVID-19, those in disadvantaged communities are less likely to get tested. The investigators are collaborating with community partners in Cumberland County, Maine to implement a public health intervention focused on making COVID-19 testing more accessible to underserved populations. The intervention includes a one-time in-person training on how to take an at-home COVID-19 test and then provision of at-home COVID-19 testing kits to make testing more accessible. Five testing kits are provided at the time of training and then provided every two months for a year, for a total of 35 testing kits.

In this study, the investigators will evaluate the impact of the at-home testing kit intervention on COVID-19 testing behavior, knowledge and attitudes. The investigators will accomplish this aim by following a community cohort, with a goal of recruiting 150 participants - 15 participants from each of our 10 population groups of interest (three groups that access different health services for low-income/uninsured, unhoused individuals, and six different immigrant groups). The investigators will administer surveys to the cohort participants every month over a 12 month period. Every month the survey will ask about testing behavior, and every other month the survey will also ask about knowledge and attitudes towards testing. In order to ensure access to COVID-19 tests, the cohort participants will be provided at-home testing kits throughout the course of the study. The primary outcome of interest is "recommended testing behavior," which is defined as taking a rapid COVID-19 test when experiencing symptoms of COVID-19 or after a close contact exposure.

The investigators hypothesize that knowledge about testing, favorable attitudes towards testing, and recommended testing behavior will increase as a result of participation in the study.

ELIGIBILITY:
Inclusion criteria:

* Individual accesses services from one of these three public health facilities - community free clinic, needle exchange program, or STD clinic
* Individual is currently unhoused or living in a Housing First development
* Individual immigrated to the US, primarily from one of these six country groups - Somalia, Angola, Iraq or Syria, Burundi or Rwanda, Democratic Republic of the Congo, or a country in Latin America

Exclusion criteria:

• Individual is <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Fairfield, MD, DrPH, Principal Investigator — MaineHealth
Locations (3):
- United States (3):
  - Greater Portland Health, Portland, Maine
  - Portland Community Free Clinic, Portland, Maine
  - Preble Street Learning Collaborative, Portland, Maine

REFERENCES:
- [Background] Clark E, Fredricks K, Woc-Colburn L, Bottazzi ME, Weatherhead J. Disproportionate impact of the COVID-19 pandemic on immigrant communities in the United States. PLoS Negl Trop Dis. 2020 Jul 13;14(7):e0008484. doi: 10.1371/journal.pntd.0008484. eCollection 2020 Jul. No abstract available. PMID 32658925
- [Background] Laurencin CT, McClinton A. The COVID-19 Pandemic: a Call to Action to Identify and Address Racial and Ethnic Disparities. J Racial Ethn Health Disparities. 2020 Jun;7(3):398-402. doi: 10.1007/s40615-020-00756-0. Epub 2020 Apr 18. PMID 32306369
- [Background] Nayak A, Islam SJ, Mehta A, Ko YA, Patel SA, Goyal A, Sullivan S, Lewis TT, Vaccarino V, Morris AA, Quyyumi AA. Impact of Social Vulnerability on COVID-19 Incidence and Outcomes in the United States. medRxiv [Preprint]. 2020 Apr 17:2020.04.10.20060962. doi: 10.1101/2020.04.10.20060962. PMID 32511437
- [Background] Price-Haywood EG, Burton J, Fort D, Seoane L. Hospitalization and Mortality among Black Patients and White Patients with Covid-19. N Engl J Med. 2020 Jun 25;382(26):2534-2543. doi: 10.1056/NEJMsa2011686. Epub 2020 May 27. PMID 32459916
- [Background] Sy KTL, Martinez ME, Rader B, White LF. Socioeconomic Disparities in Subway Use and COVID-19 Outcomes in New York City. Am J Epidemiol. 2021 Jul 1;190(7):1234-1242. doi: 10.1093/aje/kwaa277. PMID 33372209
- [Background] Moore JT, Ricaldi JN, Rose CE, Fuld J, Parise M, Kang GJ, Driscoll AK, Norris T, Wilson N, Rainisch G, Valverde E, Beresovsky V, Agnew Brune C, Oussayef NL, Rose DA, Adams LE, Awel S, Villanueva J, Meaney-Delman D, Honein MA; COVID-19 State, Tribal, Local, and Territorial Response Team. Disparities in Incidence of COVID-19 Among Underrepresented Racial/Ethnic Groups in Counties Identified as Hotspots During June 5-18, 2020 - 22 States, February-June 2020. MMWR Morb Mortal Wkly Rep. 2020 Aug 21;69(33):1122-1126. doi: 10.15585/mmwr.mm6933e1. PMID 32817602
- [Background] Millett GA, Jones AT, Benkeser D, Baral S, Mercer L, Beyrer C, Honermann B, Lankiewicz E, Mena L, Crowley JS, Sherwood J, Sullivan PS. Assessing differential impacts of COVID-19 on black communities. Ann Epidemiol. 2020 Jul;47:37-44. doi: 10.1016/j.annepidem.2020.05.003. Epub 2020 May 14. PMID 32419766

RESULTS

PARTICIPANT FLOW:
Groups:
- COVID-19 Testing: The cohort participants will attend an in-person training on how to take an at-home COVID-19 test and also be provided with five at-home test kits at the training and every other month for a total of 35 kits over the course of a year.
  Public Health Intervention Package: The intervention package consists of two components:
  1. At the time of study enrollment, participants will attend an in-person training on how to properly take an at-home COVID-19 test. Study staff will verbally walk through the steps of the test with the participant while the participant administers the test on themselves, with the opportunity to ask questions and receive corrective feedback, as needed.
  2. To make COVID-19 testing more accessible, participants will be provided five at-home COVID-19 testing kits at the training and then every other month throughout the course of the year-long study for a total of 35 kits.
Period: Overall Study
Arm/Group | COVID-19 Testing
Started | 102
Completed | 93
Not Completed | 9
Not completed — Death | 1
Not completed — Medical issues impacted ability to participate | 2
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Participants completed an enrollment survey and then were asked to complete a COVID-19 testing survey every 4 weeks for one year. All participants who completed their enrollment survey are included in this baseline analysis table (i.e. it is not dependent on how many COVID-19 testing surveys they completed).
Arm/Group | COVID-19 Testing
Number analyzed (Participants) | 93
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.5 (15)
Age, Customized [Count of Participants; unit: Participants]
  18-24 years | 7
  25-39 years | 33
  40-59 years | 34
  60 years or older | 19
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 50
  Male | 42
  Non-binary | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 45
  Black/African-American | 34
  Hispanic | 5
  Asian | 3
  Native American | 1
  Other | 2
  Not reported | 3
Region of Enrollment [Number; unit: participants] — All participants were enrolled in Portland, ME, USA
  participants
    United States | 93
Received COVID-19 vaccine [Count of Participants; unit: Participants] — Received at least 1 dose of a COVID-19 vaccine
  Participants | 84
Education level [Count of Participants; unit: Participants]
  8th grade or less | 5
  Some/all high school | 28
  Some college/technical degree/vocational | 22
  Bachelor's degree or higher | 36
  Prefer not to answer | 2
Self-reported health [Count of Participants; unit: Participants]
  Excellent | 16
  Very good | 31
  Good | 28
  Fair | 15
  Poor | 3
Employed currently [Count of Participants; unit: Participants] | 42
Health insurance [Count of Participants; unit: Participants]
  Private | 27
  Public (Medicare, Medicaid, Tricare) | 45
  Uninsured | 17
  Don't know | 4
Immigrant [Count of Participants; unit: Participants] | 39
Low income by federal poverty guidelines [Count of Participants; unit: Participants] | 51
Unhoused or history of chronic homelessness [Count of Participants; unit: Participants] | 30
Self-reported substance use [Count of Participants; unit: Participants] | 28

OUTCOME MEASURES:

1. Primary Outcome: Recommended Testing Proportion
Description: Primary outcome measures how many times a participant tested out of the total number of times they should have tested based on public health recommendations (i.e. symptomatic and/or had close contact exposure). Participants are sent a survey every month over the course of 12 months. The participant is asked if, in the past month, they had been in close contact with someone with COVID-19 and/or experienced COVID-19 symptoms. The survey then asks the participant to self-report on whether or not they took an at-home COVID-19 rapid antigen test. The data from all 12 surveys is summed to calculate a single value for "recommended testing proportion" for each participant.
  Metric = total # of times participant took COVID-19 rapid test when recommended / total # of times participant should have taken COVID-19 rapid test when recommended e.g. participant tested 7 times in total / 10 times in total when participant should have tested = 0.70 recommended testing across the 12 month time frame
Time Frame: 12 months
Population: Only 84 of the 93 participants reported an incident in at least one of their surveys that should have prompted COVID-19 testing (i.e. symptoms or exposure); therefore, only 84 participants are included in the analysis of testing behavior. Here we report the average recommended testing proportion among all 84 participants (e.g. participants on average tested 66% of the times they should have done so, according to CDC guidelines)
Measure: Mean (Standard Deviation); unit: proportion of times tested asrecommended
Arm/Group | COVID-19 Testing
Number analyzed (Participants) | 84
proportion of times tested asrecommended | 0.66 (0.29)

2. Secondary Outcome: 1) Confidence in Ability to Use COVID-19 Tests
Description: The secondary outcome measures will include various knowledge and attitude questions that capture the participants' perceptions towards COVID-19 testing. These questions have 5-pt Likert response options. Participants will answer COVID-19 testing knowledge and attitude questions at the time of enrollment and then answer the same questions every 2 months over the course of 12 months for a total of 7 time points. We will calculate an average across the responses for each item during this 12 month period.
  Metric = Average testing perception for each knowledge/attitude item
  Item 1: How confident are you in your ability to properly conduct an at-home COVID-19 test? 1 = Not confident; 2 = A little confident; 3 = Confident; 4 = Quite confident; 5 = Very confident
  *Higher score is desired (i.e. indicates greater confidence)
Time Frame: 12 months
Population: Out of the 93 enrolled participants, 1 participant never completed a survey with this item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COVID-19 Testing
Number analyzed (Participants) | 92
units on a scale | 4.16 (0.78)

3. Secondary Outcome: 2) Perceived Severity of Illness From COVID-19
Description: The secondary outcome measures will include various knowledge and attitude questions that capture the participants' perceptions towards COVID-19 testing. These questions have 5-pt Likert response options. Participants will answer COVID-19 testing knowledge and attitude questions at the time of enrollment and then answer the same questions every 2 months over the course of 12 months for a total of 7 time points. We will calculate an average across the responses for each item during this 12 month time period.
  Metric = Average testing perception for each knowledge/attitude item
  Item 2: Imagine you test positive for COVID-19. How severely do you think your health would be impacted? 1 = Not severe; 2 = A little severe; 3 = Severe; 4 = Quite severe; 5 = Very severe
  *Higher score is desired (i.e. indicates greater perceived severity around COVID illness)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COVID-19 Testing
Number analyzed (Participants) | 84
units on a scale | 2.15 (0.89)

4. Secondary Outcome: 3) Perceived Usefulness of COVID-19 Testing
Description: The secondary outcome measures will include various knowledge and attitude questions that capture the participants' perceptions towards COVID-19 testing. These questions have 5-pt Likert response options. Participants will answer COVID-19 testing knowledge and attitude questions at the time of enrollment and then answer the same questions every 2 months over the course of 12 months for a total of 7 time points. We will calculate an average across the responses for each item during this 12 month time period.
  Metric = Average testing perception for each knowledge/attitude item
  Item 3: Composite of two questions How important is it to you that you get tested for COVID-19 when you are experiencing symptoms or had a close contact?
  1 = Not important; 5 = Very important How useful do you think it is to take a COVID-19 test when you are experiencing symptoms or had a close contact?
  1 = Not at all useful; 5 = Very useful
  *Higher score is desired
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COVID-19 Testing
Number analyzed (Participants) | 84
units on a scale | 4.12 (1.02)

5. Secondary Outcome: 4) Norms Around COVID-19 Testing
Description: Secondary outcomes include various knowledge and attitude questions that capture the participants' perceptions towards COVID-19 testing. These questions have 5-pt Likert response options. Participants will answer COVID-19 testing knowledge and attitude questions at the time of enrollment and then answer the same questions every 2 months over the course of 12 months for a total of 7 time points. We will calculate an average across the responses for each item during this 12 month period.
  Metric = Average testing perception for each knowledge/attitude item
  Item 4: Combines two questions Among the people you know, how many take a COVID-19 test when they are experiencing symptoms or had a close contact?
  1 = (Almost) none of them; 5 = (Almost) all of them Overall, among the people who are important to you, how much do they approve or disapprove of taking a COVID-19 test when you have symptoms or a close contact?
  1 = disapprove a lot; 5 = approve a lot
  *Higher score is desired
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COVID-19 Testing
Number analyzed (Participants) | 84
units on a scale | 2.78 (0.92)

6. Secondary Outcome: 5) Commitment to COVID-19 Testing
Description: The secondary outcome measures will include various knowledge and attitude questions that capture the participants' perceptions towards COVID-19 testing. These questions have 5-pt Likert response options. Participants will answer COVID-19 testing knowledge and attitude questions at the time of enrollment and then answer the same questions every 2 months over the course of 12 months for a total of 7 time points. We will calculate an average across the responses for each item during this 12 month time period.
  Metric = Average testing perception for each knowledge/attitude item
  Item 5: How committed are you to taking a COVID-19 test when you are experiencing symptoms or had a close contact? 1 = Not at all committed; 2 = Somewhat committed; 3 = Committed; 4 = Quite committed; 5 = Very committed
  *Higher score is desired (i.e. indicates greater commitment towards testing)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COVID-19 Testing
Number analyzed (Participants) | 84
units on a scale | 4.05 (0.83)

ADVERSE EVENTS:
Time Frame: Adverse events were tracked for 12 months (the duration of time each participant was enrolled in the study from baseline to the final survey at the 12 month mark).
Arm/Group | COVID-19 Testing
All-Cause Mortality (participants affected / at risk) | 1/102
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 0/102

LIMITATIONS AND CAVEATS:
A major limitation was that all participants received the at-home COVID-19 tests; therefore, there was no control group for direct comparison. This approach helped facilitate research engagement among a population traditionally underrepresented in biomedical research, by allowing all participants to engage with the testing program. However, further study with a control group is needed to determine the true effect of this at-home testing program on desired testing behavior in these populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT05270694/Prot_SAP_ICF_000.pdf